CLINICAL TRIAL: NCT03718533
Title: The ELTION Study - A Multicenter Open-label Interventional Study of Eltrombopag in Patients With Poor Graft Function After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Study of Efficacy and Safety of Eltrombopag in Patients With Poor Graft Function
Acronym: ELTION
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In the context of COVID-19 pandemic, the benefit / risk ratio of the participation of a patient with pancytopenia could be compromised. The decision of this premature termination was not the consequence of any safety reason inherent to the drug.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CETB115EES03; 2018-001129-15 (EudraCT Number)
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Poor Graft Function
Keywords: Eltrombopag; Hematological response; Poor graft function; Stem cell transplantation; Adult; ELTION; Phase II
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Patients received eltrombopag orally once daily up to 36 weeks.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag was provided as 50 mg or 25 mg film-coated tablets for oral use administration

SUMMARY:
The purpose of this study was to evaluate the efficacy of eltrombopag for poor graft function (PGF) on overall hematologic response (partial and complete), as determined by platelet, hemoglobin and neutrophil counts by 16 weeks after the initiation of eltrombopag in patients with poor graft function after allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
This was an open-label, single-arm phase II study, in which participants diagnosed with PGF after allo-HSCT were treated with eltrombopag up to week 36 or until the participant's premature withdrawal.

The study consisted of the following periods:

* Screening Period (baseline): the participant screening criteria was reviewed, and the procedures established in the evaluation schedule were performed.
* Treatment Period: from administration of the first dose of eltrombopag until time when participant permanently stopped taking study treatment for any reason or until 36 weeks had passed. Eltrombopag was initiated on Day 1 at a dose of 150 mg once daily (75 mg daily in Asian ancestry participants). During the Treatment Period, participants were evaluated weekly during the first month, every 2 weeks during the next 2 months and subsequently every 4 weeks until week 24. For the last 3 months, participants were followed every 6 weeks Only participants who had a partial or complete response at Week 16 continued to receive eltrombopag up to Week 36 or until loss of response (defined as a decrease in blood counts to levels that did not continue to meet the criteria for response established in the protocol), unacceptable toxicity, or discontinuation for any other reason.

Participants who discontinued eltrombopag because efficacy, continued in the study and attended the scheduled visits of Treatment Period as per protocol. If loss of response occurred, eltrombopag was reintroduced at the last effective dose.

* Final Visit (or Early Withdrawal): this visit took place 30 days after completion of the Treatment Period, or premature participant withdrawal.
* Follow-up for Survival: all participants who discontinued from the study, regardless the reason of discontinuation, were followed for survival for 24 and 36 weeks, unless they withdrew their consent, died or were lost-to follow-up, in which case study visits were no longer carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be able to understand and communicate with the investigator and comply with the requirements of the study and must provide written, signed and dated informed consent form before any study assessment is performed
2. Male of female patients ≥ 18 years of age
3. Patients diagnosed with primary or secondary poor graft function (PGF) defined as two or more cytopenias after day +30 post-transplant (re-tested in a peripheral blood analysis at screening):

   1. Platelet count <20,000/ µL (mandatory)
   2. Absolute neutrophil count (ANC) <1,000/µL
   3. Hemoglobin <100 g/L
4. Presence of donor chimerism >90% in screening visit
5. Karnofsky status ≥90% (Karnofsky assessment must be performed within 7 days prior to Day 1)

Exclusion Criteria:

1. Pregnant or nursing (lactating women).
2. Evidence of active acute or chronic graft versus host disease (GVHD).
3. Evidence of any active malignancy.
4. Subjects who are human immune deficiency virus (HIV), hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg) positive in screening visit.
5. Cytogenetic abnormality in chromosome 7 present before the allo-HSC.
6. Evidence of any clonal abnormality on cytogenetics (in bone marrow analysis).

   * A local post-transplant conventional cytogenetic assessment should be available within 8 weeks before Day 1.
   * If the cytogenetics is not valuable, i.e, it does not show metaphases, a FISH for MDS-related most frequent abnormalities including chromosome 7 is accepted.

   As a consequence, patients with dry tap bone marrow aspiration are NOT eligible.
7. Evidence of bone marrow involvement or progression of the underlying disease assessed by the applicable methods in each case.
8. Evidence of thrombotic microangiopathy.
9. Evidence of possible causes of cytopenia other than PGF (active infections, myelotoxic drugs, hypersplenism…).
10. Prior use of any thrombopoietin receptor (TPO-R) agonists for PGF.
11. AST or ALT levels >3 x ULN.
12. Creatinine level ≥1.5 x ULN.
13. Total bilirubin level ≥1.5 x ULN.
14. Previous thromboembolic event (other than line-related upper extremity thrombosis)
15. Hypersensitivity to eltrombopag or its components.
16. Clinically significant ECG abnormality history or current diagnosis of cardiac disease indicating significant risk of safety for subjects participating in the study such as uncontrolled or significant cardiac disease or impaired cardiac function including any of the following:

    1. . Corrected QTc > 450 msec (male subjects), > 460 msec (female subjects) using Fredericia correction (QTcF) on the screening ECG
    2. . Myocardial infarction
    3. . Uncontrolled congestive heart failure
    4. . Unstable angina
    5. . Congenital long QT syndrome.
17. Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment.
18. Patient with liver cirrhosis.
19. Risk factors for Torsade de Pointes including uncorrected hypokalemia or hypomagnesemia.
20. Subjects with any serious and/ or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with patient´s safety, obtaining informed consent or compliance with the study procedures as per investigator discretion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Plain Language Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 7 centers in 1 country (Spain).
Pre-assignment Details: A total of 25 participants were screened in this study of which 15 failed screening and 10 participants were enrolled in the study.
Groups:
- Eltrombopag: Participants received eltrombopag orally once daily up to 36 weeks.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 10
Completed | 3
Not Completed | 7
Not completed — Myelodysplastic syndrome and study indication | 1
Not completed — Protocol deviation | 1
Not completed — Disease progression | 1
Not completed — Relapse | 1
Not completed — Physician Decision | 2
Not completed — Physician Decision and Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: Years] | 52.5 [23.0 to 72.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9
  Native American | 1

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response Rate by 16 Weeks After the Initiation of Eltrombopag
Description: Hematologic response rate was defined as the percentage of participants who met the criteria of either complete response (CR) or partial response (PR) by Week 16. PR was defined when any of the following: Platelet count ≥ 20000/microliter(μL) (with platelet transfusion independence), absolute neutrophil count (ANC) ≥1000/μL (when pretreatment ANC was <1000/μL) and/or hemoglobin (Hb) ≥100 gram(g)/ liter(L) (when pretreatment Hb was <100g/L) (with red blood cells transfusion independence), confirmed in two blood tests separated a minimum of 7 days. CR was defined when all of the following: platelet count ≥100000/μL, ANC ≥1500/μL (when pretreatment ANC was <1000/μL) and Hb ≥110 g/L (when pretreatment Hb was <100g/L), confirmed in two blood tests separated a minimum of 7 days. Participants who discontinued before Week 16 were considered as responders if, in the last evaluation, they had PR or CR. The 95% Confidence Interval (CI) was the binomial exact CI based on Clopper-Pearson method.
Time Frame: Baseline up to Week 16
Population: All participants to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Percentage of participants | 40.0 [12.2 to 73.8]

2. Secondary Outcome: Percentage of Participants Who Had a Response in the Neutrophil Lineage
Description: Percentage of participants who had a response (partial or complete) in the neutrophil lineage. A partial response in the neutrophil lineage was defined as absolute neutrophil count (ANC) ≥1000/ µL (when pretreatment ANC was <1000/μL) confirmed in two consecutive blood tests separated a minimum of 7 days. A complete response in the neutrophil lineage was defined as ANC ≥ 1500/ µL (when pretreatment ANC was <1000/μL) confirmed in two consecutive blood tests separated a minimum of 7 days. The 95% CI was the binomial exact CI based on Clopper-Pearson method
Time Frame: Week 16, 20, 24, 30 and 36
Population: All participants to whom study treatment was assigned and pretreatment ANC was <1000 µL. Number analyzed signified number of participants that reached the study week.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 4
Percentage of Participants
  Week 16: number analyzed (Participants) | 1
  Week 16 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=1) had a response
  Week 20: number analyzed (Participants) | 1
  Week 20 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=1) had a response
  Week 24: number analyzed (Participants) | 1
  Week 24 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=1) had a response
  Week 30: number analyzed (Participants) | 1
  Week 30 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=1) had a response
  Week 36: number analyzed (Participants) | 1
  Week 36 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=1) had a response

3. Secondary Outcome: Percentage of Participants Who Had a Response in the Platelet Lineage
Description: Percentage of participants who had a response (partial or complete) in the platelet lineage. A partial response in the platelet lineage was defined as platelet count ≥20000/µL (with platelet transfusion independence) confirmed in two consecutive blood tests separated a minimum of 7 days. A complete response in the platelet lineage was defined as platelet count ≥ 100000/µL confirmed in two consecutive blood tests separated a minimum of 7 days. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: Week 16, 20, 24, 30 and 36
Population: All participants to whom study treatment was assigned. Number analyzed signified number of participants that reached the study week.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Percentage of participants
  Week 16: number analyzed (Participants) | 6
  Week 16 | 66.7 [22.3 to 95.7]
  Week 20: number analyzed (Participants) | 6
  Week 20 | 66.7 [22.3 to 95.7]
  Week 24: number analyzed (Participants) | 6
  Week 24 | 83.3 [35.9 to 99.6]
  Week 30: number analyzed (Participants) | 5
  Week 30 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=5) had a response
  Week 36: number analyzed (Participants) | 3
  Week 36 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=3) had a response

4. Secondary Outcome: Percentage of Participants Who Had a Response in the Hemoglobin Lineage
Description: Percentage of participants who had a response (partial or complete) in the hemoglobin (Hb) lineage. A partial response in the Hb lineage was defined as Hb ≥100 g/L (when pretreatment Hb was <100g/L) (with RBC transfusion independence), confirmed in two consecutive blood tests separated a minimum of 7 days. A complete response in the Hb lineage was defined as Hb≥ 110 g/L (when pretreatment Hb was <100g/L) confirmed in two consecutive blood tests separated a minimum of 7 days. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: Week 16, 20, 24, 30 and 36
Population: All participants to whom study treatment was assigned and pretreatment Hb <100g/L. Number analyzed signified number of participants that reached the study week.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 6
Percentage of participants
  Week 16: number analyzed (Participants) | 5
  Week 16 | 60.0 [14.7 to 94.7]
  Week 20: number analyzed (Participants) | 5
  Week 20 | 60.0 [14.7 to 94.7]
  Week 24: number analyzed (Participants) | 5
  Week 24 | 80.0 [28.4 to 99.5]
  Week 30: number analyzed (Participants) | 4
  Week 30 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=4) had a response
  Week 36: number analyzed (Participants) | 2
  Week 36 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=2) had a response

5. Secondary Outcome: Hematologic Response Rate at Week 24 and 36
Description: Hematologic response rate was defined as the percentage of participants who met the criteria of either complete response (CR) or partial response (PR) at 24 weeks and 36 weeks after the initiation of eltrombopag. PR was defined when any of the following: Platelet count ≥20000/microliter (μL) (with platelet transfusion independence), absolute neutrophil count (ANC) ≥1000/μL (when pretreatment ANC was <1000/μL) and/or hemoglobin (Hb) ≥100 gram (g)/ liter (L) (when pretreatment Hb was <100g/L) (with red blood cells transfusion independence), confirmed in two blood tests separated a minimum of 7 days. CR was defined when all three of the following: platelet count ≥100000/μL, ANC ≥1500/μL (when pretreatment ANC was <1000/μL) and Hb ≥110 g/L (when pretreatment Hb was <100g/L), confirmed in two blood tests separated a minimum of 7 days. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: Week 24 and 36
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Percentage of participants
  Week 24: number analyzed (Participants) | 6
  Week 24 | 83.3 [35.9 to 99.6]
  Week 36: number analyzed (Participants) | 3
  Week 36 | 100 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated as all participants analyzed (n=3) had a response

6. Secondary Outcome: Percentage of Participants Who Were Previously Platelet Transfusion-dependent and Did no Longer Require Platelet Transfusions After the Initiation of Eltrombopag
Description: Percentage of participants who received at least one platelet transfusion before starting treatment and who did no longer require platelet transfusion before and after the first 16 weeks of treatment. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: From start of treatment to end of treatment, assessed up to 36 weeks
Population: All participants to whom study treatment was assigned and who received at least one platelet transfusion before starting treatment. Number analyzed signified number of participants with evaluable data for this outcome measure at specified time points
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 7
Percentage of participants
  From start of treatment to Week 16 | 0 [NA to NA] — Not Applicable (NA) indicates confidence interval could not be calculated as no participants had platelet transfusion independence during this period
  From Week 16 to end of treatment: number analyzed (Participants) | 3
  From Week 16 to end of treatment | 66.7 [9.4 to 99.2]

7. Secondary Outcome: Percentage of Participants Who Were Previously Red Blood Cells Transfusion-dependent and Did no Longer Require Red Blood Cells Transfusions
Description: Percentage of participants who received at least one red blood cells transfusion before starting treatment and who did no longer require red blood cells transfusion before and after the first 16 weeks of treatment. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: From start of treatment to end of treatment, assessed up to 36 weeks
Population: All participants to whom study treatment was assigned and who received at least one red blood cells transfusion before starting treatment. Number analyzed signified number of participants with evaluable data for this outcome measure at specified time points
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 6
Percentage of participants
  From start of treatment to Week 16 | 16.7 [0.42 to 64.1]
  From Week 16 to end of treatment: number analyzed (Participants) | 2
  From Week 16 to end of treatment | 50 [1.2 to 98.7]

8. Secondary Outcome: Duration of Transfusion Independence
Description: Duration of transfusion independence defined as the period of time where participants did not receive any platelet or red blood cells transfusions during the treatment period
Time Frame: From start of treatment to end of treatment, assessed up to 36 weeks
Population: All participants to whom study treatment was assigned.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Days | 137.7 (110.4)

9. Secondary Outcome: Percentage of Participants Who Discontinued or Reduced the Use of Concomitant Erythropoietin (EPO) Therapy
Description: Percentage of participants who discontinued or reduced by ≥50% from baseline the use of concomitant EPO therapy while receiving eltrombopag. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: From start of treatment to end of treatment, assessed up to Week 36
Population: All participants to whom study treatment was assigned with evaluable data for this outcome measure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 8
Percentage of participants
  Discontinued EPO therapy | 37.5 [8.5 to 75.5]
  Reduced by 50% EPO therapy | 0 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated because no participants reduced by 50% EPO therapy

10. Secondary Outcome: Percentage of Participants Who Discontinued or Reduced the Use of Concomitant Granulocyte Colony-stimulating Factor (G-CSF) Therapy
Description: Percentage of participants who discontinued or reduced by ≥50% from baseline the use of concomitant G-CSF therapy while receiving eltrombopag. The 95% CI was the binomial exact CI based on Clopper-Pearson method.
Time Frame: From start of treatment to end of treatment, assessed up to Week 36
Population: All participants to whom study treatment was assigned with evaluable data for this outcome measure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 7
Percentage of participants
  Discontinued G-CSF therapy | 85.7 [42.1 to 99.7]
  Reduced by 50% G-CSF therapy | 0 [NA to NA] — Not applicable (NA) indicates confidence interval could not be calculated because no participants reduced by 50% G-CSF therapy

11. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from the date of inclusion until the date of death due to any cause was calculated using Kaplan-Meier estimated. All patients who discontinued from the study, regardless the reason of discontinuation, were followed for survival, unless they withdrew their consent, died or were lost-to follow-up, in which case were censored at the last contact.
Time Frame: From start of treatment until the date of death, assessed up to 40 weeks
Population: All participants to whom study treatment was assigned.
Measure: Median (Standard Error); unit: Weeks
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Weeks | NA (NA) — Not applicable (NA) indicates median OS was not reached

12. Secondary Outcome: Overall Survival Rate at 24 and 36 Weeks
Description: Overall survival rate defined as the rate estimate of the percentage of participants who were alive at 24 and 36 weeks. All patients who discontinued from the study, regardless the reason of discontinuation, were followed for survival at Week 24 and 36, unless they withdrew their consent, died or were lost-to follow-up, in which case were censored at the last contact.
Time Frame: Week 24 and 36
Population: All participants to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Percentage of participants
  Week 24 | 90.0 [71.4 to 100.0]
  Week 36 | 80.0 [52.5 to 100.0]

13. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths due to any cause were collected from first dose of study medication to 30 days after the last dose of eltrombopag. Post-treament survival follow-up deaths were collected from day 31 after last dose of study medication to end of study.
  Participants who completed treatment with study drug as planned at Week 36, were followed up until Week 40 and deaths that occurred within that time frame were counted as on-treatment. For all participants who discontinued from eltrombopag, post-treatment deaths due to any cause were collected after the on-treatment period until end of survival follow-up period.
Time Frame: On-treatment deaths: Up to 40 weeks. Post-treatment survival follow-up deaths: up to 40 weeks
Population: All participants to whom study treatment was assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 10
Participants
  On-treatment deaths | 0
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 7
  Post-treatment survival follow-up deaths | 2
  All deaths | 2

ADVERSE EVENTS:
Time Frame: From day of first dose of study medication to the last dose of study medication plus 30 days, up to 40 weeks. Deaths were collected in the post treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to 40 weeks. These are not considered AEs
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period.
Groups:
- Eltrombopag (On-treatment): AEs during on-treatment period (up to 30 days post-treatment)
- Eltrombopag (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Eltrombopag (On-treatment) | Eltrombopag (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 0/10 | 2/7
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/0
Other Adverse Events (participants affected / at risk) | 10/10 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (On-treatment) (N=10) | Eltrombopag (Post-treatment Survival Follow-up) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | NA
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | NA
Chimerism (Congenital, familial and genetic disorders) | 1 (1) | NA
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 (1) | NA
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | NA
Pyrexia (General disorders) | 1 (3) | NA
Urosepsis (Infections and infestations) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (On-treatment) (N=10) | Eltrombopag (Post-treatment Survival Follow-up) (N=0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | NA
Headache (Nervous system disorders) | 1 (1) | NA
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 4 (5) | NA
Asthenia (General disorders) | 3 (3) | NA
Hypogammaglobulinaemia (Immune system disorders) | 1 (3) | NA
Influenza (Infections and infestations) | 1 (1) | NA
Iron overload (Metabolism and nutrition disorders) | 2 (2) | NA
Nasopharyngitis (Infections and infestations) | 2 (2) | NA
Oral candidiasis (Infections and infestations) | 1 (1) | NA
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | NA
Breast operation (Surgical and medical procedures) | 1 (1) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA
Cytomegalovirus infection (Infections and infestations) | 1 (1) | NA
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 (1) | NA
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | NA
Papiloma excision (Surgical and medical procedures) | 1 (1) | NA
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | NA
Anaemia (Blood and lymphatic system disorders) | 1 (1) | NA
Finger amputation (Surgical and medical procedures) | 1 (1) | NA
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | NA
Upper respiratory tract infection (Infections and infestations) | 2 (2) | NA
Urine analysis abnormal (Investigations) | 1 (1) | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Dizziness (Nervous system disorders) | 1 (1) | NA
Eye pruritus (Eye disorders) | 1 (1) | NA
Neutrophil count decreased (Investigations) | 1 (1) | NA
Oedema peripheral (General disorders) | 1 (1) | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Clostridium test positive (Investigations) | 1 (1) | NA
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT03718533/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT03718533/SAP_001.pdf